CLINICAL TRIAL: NCT04014192
Title: Effects of SGLT2 Inhibitors on Islet Cell Function and Insulin Sensitivity in Patients of Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yuan-SGLT2
Record Dates: First submitted 2019-07-07; First posted 2019-07-10 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Sodium and Glucose Synergistic Transporter 2 Inhibitor; Beta Cell Function; Alpha Cell Function; Insulin Sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — dapagliflozin; empagliflozin; Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dapagliflozin Group (Experimental): 10mg/d for one week
  Interventions: Drug: Dapagliflozin
- Empagliflozin Group (Experimental): 10mg/d for one week
  Interventions: Drug: Empagliflozin
- Canagliflozin Group (Experimental): 100mg/d for one week
  Interventions: Drug: Canagliflozin
- Normal Glucose Tolerance Group (No Intervention)

INTERVENTIONS:
Drug: Dapagliflozin — Treated with dapagliflozin 10mg/d for one week.
  Arms: Dapagliflozin Group
Drug: Empagliflozin — Treated with empagliflozin 10mg/d for one week.
  Arms: Empagliflozin Group
Drug: Canagliflozin — Treated with canagliflozin 100mg/d for one week.
  Arms: Canagliflozin Group

SUMMARY:
The main pathogenesis of type 2 diabetes mellitus is insulin resistance and insufficient secretion of insulin by pancreatic beta cells. SGLT2 (sodium-glucose synergistic transporter 2) inhibitor is a kind of newly developed hypoglycemic medicine, which increases urinary glucose excretion and lowers blood glucose in an insulin-independent manner. The mechanisms of its effects on insulin resistance, insulin secretion by pancreatic beta cells and glucagon secretion by pancreatic alpha cells, are not well studied in domestic and foreign, and there is no unified conclusion. A few studies concerning SGLT2 inhibitors have observed that insulin resistance and islet beta cell secretion function can be improved by the improvement of glucotoxicity and lipotoxicity, but its effect on pancreatic alpha cell function to increase glucagon level, thereby increasing liver glucose output, may be one of the mechanisms of its side effects. In this study, patients with type 2 diabetes mellitus were treated with three domestic listed SGLT2 inhibitors (dapagliflozin, empagliflozin and canagliflozin) for one week, which were expected to improve the glucotoxicity, but excluding the effects on lipotoxicity and body weight, to observe the changes of islet beta cell and alpha cell function and insulin sensitivity. Three different SGLT2 inhibitors were used in order to make clear whether this effect is the unique effect of different structure of drugs or the similar effect of this kind of drugs.

DETAILED DESCRIPTION:
In this study, type 2 diabetes patients were treated with three kinds of SGLT2 inhibitors (dapagliflozin, empagliflozin and canagliflozin) for one week. With routine dose applied, (dapagliflozin 10mg/d, empagliflozin 10mg/d, canagliflozin 100mg/d), blood glucose level could be improved with small expected effect on body weight and no effect in lipid metabolism after the treatment period of one week. Normal glucose tolerance subjects (diagnosed of OGTT) were included as the control group.According to previous studies in three major SGLT2 inhibitors currently on the market, an increase in urinary glucose excretion and a decrease in blood glucose within three days after application in mice and human could be observed. Therefore, the short-term treatment cycle in this study is intended to be set at one week, and can be extended to two weeks if there is no significant decrease in blood glucose.

The insulin sensitivity, islet beta cell secretion function and islet alpha cell function of diabetic patients were measured at baseline (before taking SGLT2 inhibitors) and one week after taking SGLT2 inhibitors, of normal glucose tolerance subjects were measured only at baseline. The effect of SGLT2 inhibitors on islet cell function and insulin sensitivity would be evaluated in order to study the extrarenal action mechanism of SGLT2 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* (1)According to the diagnostic criteria of World Health Organization (WHO) in 1999, type 2 diabetes mellitus was diagnosed clinically. The age ranged from 18 to 70 years (including 18 and 70 years). There was no limit to the duration of diabetes mellitus and gender.
* (2)Basic antidiabetic therapy is not limited.
* (3)HbA1c ≥ 7%.
* (4)eGFR ≥60 ml/min；without contraindications to SGLT2 Inhibitors.
* (5)Sign written consent form voluntarily.

Exclusion Criteria:

* (1)Other types of diabetes mellitus.
* (2)Unstable control of blood glucose(fasting blood glucose > 11.1 mmol/L).
* (3)Acute complications of diabetes mellitus within 6 months.
* (4)History of myocardial infarction or stroke within 6 months, or existing severe cardiovascular disease and risk.
* (5)Abnormal liver function [i.e. serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is 1.5 times higher than the upper limit of normal value].
* (6)Severe hypertension that defined as systolic blood pressure ≥160 mmHg, diastolic blood pressure ≥90 mmHg with drug therapy, or hypotension (resting seat blood pressure < 90/50 mmHg).
* (7)psychosis, alcohol dependence or history of drug abuse, lactation women, participation in other studies three months before the trial, allergic constitution or allergic to a variety of drug and those researchers think inappropriate to the research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to post-treatment in insulin sensitivity. | Baseline, Week 1(extended to Week 2 if without significantly decrease in blood glucose)
  Insulin sensitivity is calculated by the following formula according to blood glucose and insulin levels in OGTT (Oral Glucose Tolerance Test).
  1.1 OGTT Matsuda and De Fronzo Insulin Sensitivity Index（ISOGTT）：10000/square root(Gluc0×Ins0×mean Gluc×mean Ins)。Mean gluc and mean Ins are average values calculated by each value in 0, 60, 120 and 180 minutes of OGTT.
  1.2 QUICKI（quantitative insulin sensitivity check index）model：1/(log[Ins0]+ log[Gluc0]) 1.3 HOMA-IR：(Gluc0×Ins0)/22.5
Change from baseline to post-treatment in islet beta cell secretory function. | Baseline, Week 1(extended to Week 2 if without significantly decrease in blood glucose)
  Islet beta cell secretory function is calculated by area under the curve of blood glucose、 insulin、C-peptide in OGTT and following formula above.
  2.1 Stumvoll first phase insulin secretion：1,194+4.724×Ins0-117.0 ×Gluc60 + 1.414×Ins60 2.2 Stumvoll second phase insulin secretion：295+0.349×Ins60-25.72×Gluc60+1.107×Ins0 2.3 HOMA-β：(20×Ins0)/(Gluc0-3.5)
Change from baseline to post-treatment in islet alpha cell secretory function. | Baseline, Week 1(extended to Week 2 if without significantly decrease in blood glucose)
  Islet Alpha Cell secretory function is calculated by area under the curve of blood glucose、glucagon level in OGTT.

SECONDARY OUTCOMES:
Change from baseline to post-treatment in weight. | Baseline, Week 1(extended to Week 2 if without significantly decrease in blood glucose)
Change from baseline to post-treatment in fasting blood glucose and non-fasting blood glucose. | Baseline, Week 1(extended to Week 2 if without significantly decrease in blood glucose)
Change from baseline to post-treatment in fasting insulin level. | Baseline, Week 1(extended to Week 2 if without significantly decrease in blood glucose)
Change from baseline to post-treatment in blood lipid including cholesterol, triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol. | Baseline, Week 1(extended to Week 2 if without significantly decrease in blood glucose)
Change from baseline to post-treatment in urine volume and urine glucose level. | Baseline, Week 1(extended to Week 2 if without significantly decrease in blood glucose)
Change from baseline to post-treatment in urinary output of uric acid, sodium, calcium, and phosphorus. | Baseline, Week 1(extended to Week 2 if without significantly decrease in blood glucose)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuan T, Liu S, Dong Y, Fu Y, Tang Y, Zhao W. Effects of dapagliflozin on serum and urinary uric acid levels in patients with type 2 diabetes: a prospective pilot trial. Diabetol Metab Syndr. 2020 Oct 27;12:92. doi: 10.1186/s13098-020-00600-9. eCollection 2020. PMID 33117454